CLINICAL TRIAL: NCT03056781
Title: Emotional Response in Psychiatric and Control Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Elizabeth A. Martin, Assistant Professor, University of California, Irvine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-2945
Record Dates: First submitted 2017-01-03; First posted 2017-02-17 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Schizophrenia; Emotions
MeSH Terms: conditions — Schizophrenia | interventions — Drug Interactions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- social interaction (Experimental): Participants will engage in a social interaction with another person
  Interventions: Behavioral: social interaction
- food consumption (Experimental): Participants will be offered food stuffs to eat/drink
  Interventions: Behavioral: food consumption

INTERVENTIONS:
Behavioral: social interaction — Participants will engage in a social interaction with another person
  Arms: social interaction
Behavioral: food consumption — Participants will be offered food stuffs to eat/drink
  Arms: food consumption

SUMMARY:
The purpose of this research is to understand how the emotions of people with different mental health concerns (e.g., people with schizophrenia, people with major depressive disorder) differ from individuals without mental health concerns. A large body of literature suggests that people with mental illnesses have emotional abnormalities compared to healthy individuals, but a number of these abnormalities are not well understood. For example, often people with schizophrenia report on questionnaires that they experience fewer pleasant emotions when talking with other people, but some evidence suggests these individuals report a similar amount of pleasant emotion when they are actually engaged in a pleasant activity. Thus, it is unclear the extent to which reports of emotional abnormalities extend to a more real-world setting. In the tasks in the current proposal, participants will engage in a series of tasks designed to assess their emotional functioning. These tasks involve viewing emotional stimuli on the computer, engaging in social interactions, and consuming small amounts of food. In all tasks, participants will make ratings of their experiences of pleasure (and displeasure). We will then compare the experiences of patient groups to those of healthy individuals to test how emotional ratings might differ across these tasks.

ELIGIBILITY:
Inclusion Criteria:

* For control participants, you are eligible to participate in this study if you are between 18 and 65 years of age, you are fluent in English, and you have not been clinically diagnosed with a psychiatric disorder.
* For psychiatric patients, you are eligible to participate in this study if you are between 18 and 65 years of age, you are fluent in English, and you have been clinically diagnosed with schizophrenia, schizoaffective disorder, or depression with no recent hospitalization or changes in your psychiatric medications.

Exclusion Criteria:

* For control participants, you are not eligible to participate in the study if you have a history of stroke or a current history of substance or alcohol dependence. You are also not eligible to participate in this study if you have had a diagnosis of substance abuse in the past three months. You are not eligible to participate if you have a current or past history of a major medical illness, significant tremors, a history of a head injury or prolonged unconsciousness.
* For psychiatric patients, you are not eligible to participate in the study if you have had major changes to your psychotropic medications within the last two months, have a history of stroke or a current history of substance or alcohol dependence. You are also not eligible to participate in this study if you have had a diagnosis of substance abuse in the past three months, a current or past history of a major medical illness, significant tremors, or a history of a head injury or prolonged unconsciousness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Social Anhedonia Scale | 1 day
  measures social anhedonia
Physical Anhedonia Scale | 1 day
  measures physical anhedonia
EEG activity | 1 day
  physiological parameter
Verbal behavioral rating | 1 day
  how many words are spoken throughout the task
Non-verbal behavioral rating | 1 day
  how many gestures are made throughout the task
International Personality Item Pool questionnaires | 1 day
  measure of personality

SECONDARY OUTCOMES:
Following Affective States test | 1 day
  questionnaire re: how much participants follow or ignore their emotions
AMNART | 1 day
  measure of verbal IQ
MMSE | 1 day
  measure of mental status

CONTACTS AND LOCATIONS:
Locations (1):
- Social Ecology 1, Irvine, California, United States